CLINICAL TRIAL: NCT06899009
Title: Ventilator Settings and Outcomes in Pediatric Patients on ECMO for Severe Respiratory Failure - a Posthoc Analysis of the ELSO Registry
Brief Title: Ventilator Settings and Outcomes in Pediatric Patients on ECMO for Severe Respiratory Failure
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: Ped.ECMO.1
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Respiratory Failure (Pediatric Patients)
Keywords: Ventilation practice; Critically ill children; Mechanical ventilation; Extracorporeal membrane oxygenation; Extracorporeal lief support
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with respiratory failure on ECMO

SUMMARY:
This study aims to describe the effects of ECMO initiation on the intensity of ventilation in the first 24 hours after ECMO initiation and to explore associations between changes in ventilation intensity and hospital mortality in critically ill pediatric patients requiring ECMO for respiratory failure, using the 'Extracorporeal Life Support Organization' (ELSO) registry.

DETAILED DESCRIPTION:
Rationale:

Despite the growing use of ECMO in critically ill pediatric patients, uncertainties remain to what extent adjustments of ventilator settings after ECMO initiation are associated with mortality.

Objectives:

1. To describe the effects of ECMO initiation on the intensity of ventilation in the first 24 hours after ECMO initiation; and
2. To explore associations between changes in ventilation intensity and hospital mortality in critically ill pediatric patients requiring ECMO for respiratory failure

Hypothesis:

1. Ventilation intensity decreases following initiation of ECMO; and
2. A decrease in ventilation intensity is associated with lower hospital mortality in critically ill pediatric patients.

Study design:

This is a posthoc analysis of the ELSO registry.

Study population:

For this analysis, data will be obtained from the ELSO registry. All pediatric patients (aged ≥29 days to ≤18 years) receiving ECMO for a pulmonary indication between January 1, 2012, and December 31, 2022 will be included. Patients with missing ventilatory variables required to assess ventilation intensity and patients lost to follow up with respect to hospital mortality will be excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (aged ≥29 days to ≤18 years) receiving ECMO between January 1, 2012, and December 31, 2022, in an ELSO affiliated center; and
2. Requiring ECMO for a pulmonary indication.

Exclusion Criteria:

1. Patients with missing ventilatory variables required to assess ventilation intensity;
2. patients who were lost to follow up with respect to hospital mortality.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Critically ill pediatric patients receiving ECMO for pulmonary indications
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | Up to 90 days of study or whatever comes first

SECONDARY OUTCOMES:
Hospital length of stay | Up to 90 days of study or whatever comes first
Duration of ECMO run | Up to 90 days of study or whatever comes first
Duration of invasive ventilation | Up to 90 days of study or whatever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Martin CJ Kneyber, MD PhD FCCM, Principal Investigator — University Medical Center Groningen; Marcus J Schultz, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Frederique Paulus, RN PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No